CLINICAL TRIAL: NCT00488891
Title: The Paliperidone ER Outcomes Study of Schizophrenia Patients in Typical Clinical Practice
Brief Title: The Paliperidone ER Observational Study of Economic, Functional, and Clinical Outcomes in Patients With Schizophrenia
Acronym: POST
Status: Terminated | Type: Observational
Why Stopped: The study was terminated because it was not enrolling at the expected rate
Sponsor: Ortho-McNeil Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR014143; PAL-OUT-003 (Other: Ortho-McNeil Janssen Scientific Affairs, LLC)
Record Dates: First submitted 2007-06-18; First posted 2007-06-20 (Estimated); Last update posted 2012-08-29 (Estimated); Status verified 2012-08

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Paliperdone ER; Invega; Observational; Antipsychotic agents
MeSH Terms: conditions — Schizophrenia | interventions — Paliperidone Palmitate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — 10 mL blood sample is collected from patients who consent to the pharmacogenomic component of the study.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Paliperidone extended release (ER): Drug: Paliperidone ER will be prescribed to the patients at the investigator's discretion. Patient receive their medication according to usual care in their treatment setting ie, no study drug is provided
  Interventions: Drug: Paliperidone ER
- Atypical antipsychotics agent (AAP): AAP includes quetiapine, risperidone, olanzapine, ziprasidone or aripiprazole. Dosage and administration of antipsychotics will be prescribed at the investigator's discretion
  Interventions: Drug: Atypical antipsychotics (AAP)

INTERVENTIONS:
Drug: Paliperidone ER — Route = oral. Paliperidone ER will be prescribed to the patients at the investigator's discretion. Patient receive their medication according to usual care in their treatment setting ie, no study drug is provided
  Other Names: Invega
  Groups: Paliperidone extended release (ER)
Drug: Atypical antipsychotics (AAP) — Route = oral. AAP including quetiapine, risperidone, olanzapine, ziprasidone or aripiprazole. Dosage and administration of antipsychotics will be prescribed at the investigator's discretion
  Groups: Atypical antipsychotics agent (AAP)

SUMMARY:
The purpose of this study is to examine the long-term economic, functional and clinical outcomes in schizophrenia patients who require a change in antipsychotic treatment, and are changed to either paliperidone extended release (ER) or another oral atypical antipsychotic agent (AAP) including aripiprazole, olanzapine, quetiapine, risperidone, or ziprasidone.

DETAILED DESCRIPTION:
This is a 12-month, retrospective (a study that looks backward in time, usually using medical records and interviews with patients who are already known to have a disease)/prospective (a study in which the patients are identified and then followed forward in time for the outcome of the study), open-label (all people involved know the identity of the assigned drug) study of clinical, functional and economic outcomes in schizophrenia patients who require a change in antipsychotic treatment. The patients will be randomly (study drug assigned by chance like flipping a coin) assigned to receive either paliperidone extended release (ER) or one of two other prescriber-selected oral atypical antipsychotic (AAPs). The AAPs include aripiprazole, olanzapine, quetiapine, risperidone, or ziprasidone. Baseline will be defined as the time when the patient begins to take paliperidone ER or the other AAP. The study has a "pre/post" design in which paliperidone ER patients serve as their own controls for the analyses of healthcare utilization. If a potential patient needs to switch from their current antipsychotic medication they are eligible for this study. The investigator will determine that the patient may benefit equally from switching to either paliperidone ER (extended release) or to either of 2 other antipsychotics. Healthcare use over the 12-month period prior to baseline (the "pre-period") will be compared to the 12-month period following the start of paliperidone ER or other AAP (the "post-period"). Data for both periods will be obtained by study investigators from enrolled patients' medical charts. Patients will continue to be followed in the study, regardless of change in treatment, until visit 5 at month 12 or if withdrawn from the study. All patients will receive medical care consistent with local medical practices.

ELIGIBILITY:
Inclusion Criteria:

* Must have a clinical diagnosis of schizophrenia for at least 1 year prior to screening
* Had been receiving treatment with antipsychotics, but is judged to be a candidate for changing antipsychotic on the basis of either persistent symptoms or continuing side effects
* Treating physician has determined, before the patient enters the study, that starting paliperidone extended release (ER) or another of at least two possible atypical antipsychotics (AAPs) is an appropriate treatment for the patient
* Likely to be managed as outpatient
* Must have signed the informed consent form for DNA pharmacogenomic

Exclusion Criteria:

* Have mental retardation, dementia, bipolar, schizoaffective disorder, schizophreniform disease, other Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV) psychiatric disorders or deteriorating neurological illnesses as determined by clinical evaluation
* Established treatment-resistant schizophrenia, defined as those who have had treatment failures with adequate trials of two second generation atypicals, previous treatment with clozapine, or 4 or more hospitalizations in the last 12 months
* History of recent violence or at immediate risk of suicide, or harming self or others, or of causing damage to property, in the judgment of the investigator
* Patients who are unable to swallow the medication whole
* History or circumstances that may increase the risk of occurrence of torsade de pointes and/or sudden death in association with the use of drugs that prolong the QTc interval, including bradycardia, hypokalemia or hypomagnesemia, concomitant use of drugs that prolong the QTc interval, or presence of congenital long QT syndrome
* Pregnant (as confirmed by urine pregnancy test performed at baseline), planning to become pregnant, or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The majority of patients with schizophrenia are treated in the outpatient setting. Therefore, this study will focus largely on the population treated in Community Mental Health Centers (CMHCs), Veteran Affairs (VAs) Centers, as well as private practice and other treatment settings.
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2007-04; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Changes in the yearly rate of hospital admissions before and after treatment with paliperidone extended release (ER) | 12 months before and post baseline
  The baseline is referred to month 0; Baseline is the time when patients are initiated on paliperidone ER or on any other oral atypical antipsychotics [AAP]).

SECONDARY OUTCOMES:
Change from baseline in Clinical Global Impression of the severity (CGI-S) scale | Baseline to Month 12
  This scale measures global severity of illness at a given point in time. Treating physician rates the severity of a patients condition on a seven-point scale ranging from 1 (no symptoms) to 7 (very severe).
Change from baseline in Positive and Negative Syndrome Scale (PANSS) | Baseline to Month 12
  This is a 30-item scale that was designed to assess various symptoms of schizophrenia including delusions, grandiosity, blunted affect, poor attention, and poor impulse control. The 30 symptoms are rated on a 7-point scale that ranges from 1 (absent) to 7 (extreme psychopathology).
Change from baseline in Personal and Social Performance Scale (PSP and SF-36) | Baseline to Month 12
  The PSP is a clinician-based rating instrument providing an overall rating of personal and social functioning in psychiatric patients on a scale of 0 (grossly impaired functioning) to 100 (excellent functioning).
Change from baseline in Independent Living Skills Survey (ILSS) | Baseline to Month 12
  It is a measure of basic functional and cognitive skills of individuals that was developed and validated for use in severe and persistent mental illness including schizophrenia. These include taking care of one's personal appearance, money, possessions, residence, and health; finding and keeping a job and interacting with others.
Change from baseline in Healthcare and Social Services Resource Utilization | Baseline to Month 12
  Resource utilization includes healthcare and social services such as inpatient and outpatient hospital use, emergency room visits, and crisis team interventions.
Relapse rate | Baseline to Month 12
  Relapse is defined as: 1) Psychiatric hospitalization due to worsening symptomatology (not for social reason) 2) Deliberate self-injury, suicidal or homicidal ideation 3) Violent behaviour resulting in clinically significant injury to another person or property damage 4) An increase in the level of psychiatric care (eg, from clinic visits to day treatment) and substantial clinical deterioration, defined as a change score of 6 ("much worse") or 7 ("very much worse") on the clinicla global impression of change scale (CGI-C).
Change from baseline in Abnormal Involuntary Movement Scale (AIMS) | Baseline and Month 12
  This is a valid and reliable method of screening for tardive dyskinesia (disorder resulting in involuntary, repetitive body movements). It measures facial, oral, extremity and trunk movements as well as the patients awareness of abnormal movements. The AIMS contains 10 items on a scale from 0 (none) to 4 (severe). In addition, there are 2 items on dental status that are answered "yes" or "no."
Change from baseline in Clinical Global Impression of change scale (CGI-C) | Month 3 to Month 12
  The CGI-C measures change from the baseline state. The treating physician assesses the patient's clinical change relative to the symptoms at baseline on a seven-point scale, ranging from 1 (very much improved) to 7 (very much worse).
Change from baseline in Short-Form 36 Health Survey (SF-36) | Baseline to Month 12
  The SF-36 is a well-validated and widely used quality of life instrument. It is a self-administered survey that measures eight domains of health including: physical functioning, role limitations due to physical health (role-physical), bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems (role-emotional) and general mental health.
Change from baseline in Medication Compliance with Antipsychotic Medication | Baseline to Month 12
  Compliance with antipsychotic medication will be documented by the investigator or designee. Compliance will be broadly categorized as always compliant, partially compliant, or never compliant.
Change from baseline in Patient Satisfaction with Antipsychotic Medication | Baseline to Month 12
  Antipsychotic Medication Satisfaction Question is assessed by a single, self-administered seven-point Likert-type question with anchor points of extremely dissatisfied, very dissatisfied, somewhat dissatisfied, neither satisfied nor dissatisfied, somewhat satisfied, very satisfied, and extremely satisfied.
Changes in safety parameters | Baseline to Month 12
  Safety parameters include treatment-emergent adverse experiences and serious adverse experiences, physical exam, monitoring of weight, vital signs, blood glucose, hemoglogin A1C, lipid panel, and regular monitoring of movement disorders via the AIMS

CONTACTS AND LOCATIONS:
Overall Officials: Ortho-McNeil Janssen Scientific Affairs, LLC Clinical Trial, Study Director — Ortho-McNeil Janssen Scientific Affairs, LLC